CLINICAL TRIAL: NCT01607229
Title: Utility of Multi-frequency Bioelectrical Impedance Compared to Deuterium Dilution for Assessment of Total Body Water
Brief Title: Multi-frequency Bioelectrical Impedance for Estimating Total Body Water by Deuterium Dilution
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Todd Schroeder, Assistant Professor of Clinical Physical Therapy, University of Southern California
Other Study IDs: BIA-D2O-TBW
Record Dates: First submitted 2012-05-08; First posted 2012-05-30 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Total Body Water Assessment
Keywords: multi-frequency; bioelectrical impedance; body composition; hydration
MeSH Terms: interventions — Observation

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- otherwise healthy with various BMI
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — no intervention used, observed measurements from 3 test devices compared to reference criterion measurement for total body water and body composition

SUMMARY:
SPECIFIC AIM:

Determine the validity of the Biospace bioelectrical impedance devices compared to deuterium water (D2O) measurements.

HYPOTHESIS:

The Biospace Body Composition Analyzers are valid tools for measuring total body water and body composition.

ELIGIBILITY:
Inclusion Criteria:

* men and women between 18-59 years of age

Exclusion Criteria:

* Acute illness (infection, recent surgery, trauma).
* pregnancy
* pacemaker or defibrillator
* We would like to standardize the procedures and measurements in the adult population first. Older adults are excluded because by including older adults at this time, we would need to increase the sample size because we believe older adults have greater fluctuations in hydration due to medications, diet, and co-morbidities.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Total Body Water differences between criterion and test devices | Baseline only
  from BIA and from D2O

SECONDARY OUTCOMES:
Total lean body mass differences between criterion and test devices | Baseline only
  From BIA and from DXA
Appendicular lean mass differences between criterion and test devices | Baseline only
  from BIA and from DXA
Trunk lean mass differences between criterion and test devices | Baseline only
  from BIA and from DXA
Total fat mass differences between criterion and test devices | Baseline only
  from BIA and from DXA

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States